CLINICAL TRIAL: NCT06208215
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Arm Study to Evaluate the Efficacy and Safety of RZ358 in Patients With Congenital Hyperinsulinism
Brief Title: RZ358 Treatment for Congenital Hyperinsulinism
Acronym: sunRIZE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rezolute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RZ358-301
Record Dates: First submitted 2023-12-06; First posted 2024-01-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Congenital Hyperinsulinism
Keywords: Hypoglycemia; Congenital Hyperinsulinism; Glucose Metabolism Disorders; Metabolic Diseases; Pancreatic Diseases; Digestive System Diseases; Hyperinsulinism
MeSH Terms: conditions — Congenital Hyperinsulinism; Hypoglycemia; Glucose Metabolism Disorders; Metabolic Diseases; Pancreatic Diseases; Digestive System Diseases; Hyperinsulinism | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- SoC (Standard-of-Care) + RZ358 (5 mg/kg) or Placebo (Placebo Comparator): Participants ≥1 year old who receive SOC therapy and 5 mg/kg of RZ358 or placebo
  Interventions: Drug: RZ358 (5 mg/kg) + SOC (Standard-of-Care) or Placebo + SOC
- SoC + RZ358 (10 mg/kg) or Placebo (Placebo Comparator): Participants ≥1 year old who receive SOC therapy and 10 mg/kg of RZ358 or placebo
  Interventions: Drug: RZ358 (10 mg/kg) or Placebo + SOC
- Open Label Arm, SoC + RZ358 (start 5mg/kg and increase to 10 mg/kg per protocol schedule (Experimental): Infant participants from ≥3 months to <1 year old who receive SOC therapy + RZ358 starting at 5 mg/kg and increasing to 10 mg/kg of RZ358, as needed, per the protocol schedule
  Interventions: Drug: RZ358 (5-10 mg/kg) + SOC

INTERVENTIONS:
Drug: RZ358 (5 mg/kg) + SOC (Standard-of-Care) or Placebo + SOC — Participants ≥1 year old who receive SOC therapy and 5 mg/kg of RZ358 or placebo
  Arms: SoC (Standard-of-Care) + RZ358 (5 mg/kg) or Placebo
Drug: RZ358 (10 mg/kg) or Placebo + SOC — Participants ≥1 year old who receive SOC therapy and 10 mg/kg of RZ358 or placebo
  Arms: SoC + RZ358 (10 mg/kg) or Placebo
Drug: RZ358 (5-10 mg/kg) + SOC — Infant participants from ≥3 months to <1 year old who receive SOC therapy + RZ358 starting at 5 mg/kg and increasing to 10 mg/kg of RZ358, as needed, per the protocol schedule
  Arms: Open Label Arm, SoC + RZ358 (start 5mg/kg and increase to 10 mg/kg per protocol schedule

SUMMARY:
The Phase 3 pivotal study is designed to evaluate the efficacy and safety of RZ358 for the treatment of congenital hyperinsulinism (HI) as add-on to standard-of-care (SOC) therapy compared to SOC alone over 24 weeks and to evaluate the longer-term safety and efficacy of RZ358 during a subsequent open-label extension (OLE) period.

DETAILED DESCRIPTION:
Congenital hyperinsulinism (HI) is the most common cause of recurrent hypoglycemia in neonates and infants with an incidence of approximately 1 in 25,000 to 1 in 50,000 live births in the general population, and as high as 1 in 2,500 in certain populations with substantial consanguinity. Despite improved recognition, there is no satisfactory treatment or cure for congenital HI. Current medical therapies for congenital HI are directed at reducing or eliminating insulin production and/or secretion from the beta-cell. These current medications, however, achieve suboptimal glycemic control and/or have undesirable side effects. A therapy which safely and effectively attenuates the activity of insulin would address an important unmet need for these and other conditions associated with HI. This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled (SOC alone), parallel-arm, efficacy, and safety study of RZ358 in participants with congenital HI who have not achieved adequate hypoglycemia control with reasonable attempts at using usual SOC medical therapy. The study will randomize approximately 48 participants (≥1 year to ≤45 years of age) in a 1:1 ratio into 2 dosing arms (5 or 10 mg/kg with) and further randomize participants within each dosing level in a 2:1 ratio to receive RZ358 as add-on to SOC or placebo as add-on to SOC. An additional open-label (OL) arm will be conducted in parallel for participants who are ≥3 months to <1 year old (n=8), Upon completion of the pivotal treatment period (24-weeks), participants may roll-over to the OLE period at the discretion of the investigator and Sponsor.

ELIGIBILITY:
Inclusion Criteria:

At screening, aged ≥ 3 months and ≤ 45 years old.

An established clinical diagnosis of congenital HI (hyperinsulinism), with or without identification of a known monogenic variant by genetic testing.

Participant has failed to achieve adequate glycemic control with appropriate and reasonable trials of locally accepted and available Standard of Care (SOC) medical therapies (e.g., diazoxide and somatostatin analogs (SSAs)) per the judgment of the investigator.

Experiencing ≥ 3 hypoglycemia events per week by screening Self-Monitoring Blood Glucose (SMBG) and average daily percent time with hypoglycemia of ≥ 8% of the monitored screening Continuous Glucose Monitor (CGM) time.

Exclusion Criteria:

Alanine aminotransaminase (ALT), aspartate aminotransaminase (AST), total bilirubin (TB), alkaline phosphatase (ALP), and gamma-glutamyl transferase (GGT) ≥ 1.5 × the upper limit of normal for the age-specific reference range, regardless of assessed significance.

Body mass index (BMI) ≥ 35 kg/m2 for participants aged 18 years and above, or BMI ≥ 99% (percentile) per Centers for Disease Control and Prevention growth charts for participants > 12 and < 18 years of age (no BMI exclusion for participants ≤ 12 years of age).

A known clinical diagnosis of diabetes or pre-diabetes, or a history of insulin dependency within 3 months of screening.

Average daily percent time with hyperglycemia ≥ 5% of the monitored screening continuous glucose monitoring (CGM) time.

Known allergy or sensitivity to RZ358 or any component of the drug.

Ages: 3 Months to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2027-11-14 (Estimated)

PRIMARY OUTCOMES:
Glycemic efficacy: Target glucose control | 24 weeks
  Change in average weekly hypoglycemia events from baseline by point-of-care Self-Monitoring Blood Glucose (SMBG)

SECONDARY OUTCOMES:
Glycemic efficacy: Occurrence of hypoglycemia | 24 weeks
  Change in average daily percent time in hypoglycemia from baseline by Continuous Glucose Monitor (CGM)
Safety Assessments: safety and tolerability of RZ358 in patients with congenital hyperinsulinism | 24 weeks, plus up to two years of Open-Label Extension (OLE) period
  Treatment emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) captured per Common Terminology Criteria for Adverse Events (CTCAE) guidelines and coadded per Medical Dictionary for Regulatory Activities (MedDRA) will be summarized by system organ class, preferred term, and analyzed by number and percentage of events by treatment groups.
  Hepatic ultrasound: evaluated for significant structural changes (e.g. peliosis Hepatitis)
  Immunogenicity assessments: Blood samples for anti-drug antibody to RZ358 will be evaluated based on the titer, and potential neutralization effects.
  Hyperglycemia events: Will be evaluated by SMBG at thresholds of >250 mg/dL and >300 mg/dL and summarized by the treatment groups.
Safety Assessments: safety and tolerability of RZ358 in patients with congenital hyperinsulinism, Laboratory tests evaluated for significant changes from baseline by treated groups | Time Frame: 24 weeks, plus up to two years of Open-Label Extension (OLE) period
  Laboratory parameters: ALT (U/L), AST (U/L), and ALP (U/L) will be evaluated for any significant changes from baseline (>3x ULN) by treatment groups.
  Vital Signs: blood pressure (mm of Hg), heart rate (beats/minute), and respiration (rate/minute) will be evaluated for any significant changes from baseline by treatment groups.
  ECG: heart rate (beats/minute), PR (milliseconds), QTcF intervals (milliseconds) will be evaluated for any significant changes from baseline by treatment groups.
Other Glycemic efficacy: Self-Monitoring Blood Glucose (SMBG) | 24 weeks
  Proportion of participants experiencing no potentially serious hypoglycemia events by SMBG.
Other Glycemic efficacy: Self-Monitoring Blood Glucose (SMBG) Weekly Assessment | 24 weeks
  Change in average weekly incidence of potentially serious hypoglycemia events by Self-Monitoring Blood Glucose (SMBG).
Other Glycemic efficacy: Continuous Glucose Monitor (CGM) Daily Assessment | 24 weeks
  Change in average daily percent time with potentially serious hypoglycemia by Continuous Glucose Monitor (CGM).
Other Glycemic efficacy: Continuous Glucose Monitor (CGM) Overnight Assessment | 24 weeks
  Change in average 8-hour overnight percent time with hypoglycemia by CGM. Change in average daily duration (min) with hypoglycemia by CGM. Proportion of participants achieving <4% average daily time in by CGM

CONTACTS AND LOCATIONS:
Overall Officials: Gopal Saha, MD, Study Director — Rezolute
Locations (18):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
- Rezolute Investigative Site, Varna, Bulgaria, Varna, Bulgaria
- Rezolute Investigative Site, Odense, Denmark, Odense, Denmark
- France (2):
  - Rezolute Investigative Site, Bron, France, Bron
  - Rezolute Investigative Site, Paris, France, Paris
- Rezolute Investigative Site, Tbilisi, Georgia, Tbilisi, Georgia
- Germany (2):
  - Rezolute Investigative Site, Berlin, Germany, Berlin
  - Rezolute Investigative Site, Dusseldorf, Germany, Düsseldorf
- Rezolute Investigative Site, Athens, Greece, Athens, Greece
- Rezolute Investigative Site, Seeb, Oman, Seeb, Oman
- Rezolute Investigative Site, Al Rayyan, Qatar, Al Rayyan, Qatar
- Spain (2):
  - Rezolute Investigative Site, Barcelona, Spain, Barcelona
  - Rezolute Investigative Site, Sevilla, Spain, Seville
- Rezolute Investigative Site, Ankara, Turkey, Ankara, Turkey (Türkiye)
- United Kingdom (2):
  - Rezolute Investigative Site, London, United Kingdom, London
  - Rezolute Investigative Site, Manchester, United Kingdom, Manchester
- Rezolute Investigative Site, Hà Nội, Vietnam, Hà Nội, Vietnam

IPD SHARING:
Plan to Share IPD: No